CLINICAL TRIAL: NCT01679262
Title: Determination of the Optimal Size of Oropharyngeal Airway; Correlation With External Body Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2007-0407
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Ear,Nose and Throat Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optimal size of OPAs (Other)
  Interventions: Device: Guedel type color-coded OPAs

INTERVENTIONS:
Device: Guedel type color-coded OPAs — The OPAs was used four different sizes as No. 8 (80 mm, green), 9 (90 mm, yellow), 10 (100 mm, red), and 11 (110 mm, orange) in regular sequence. The curvilinear distance from the incisors to the tip of the epiglottis was measured by FOB (Olympus LF-GP; Olympus Optical Co., Tokyo, Japan) with tape marking via each size of OPAs. The distance from the distal end of OPA to the tip of the epiglottis was calculated by the difference between measured distance from the incisors to the tip of the epiglottis via each OPA by FOB and typical distance from the flange to distal end of each OPA via inside tube of OPA. When the size of OPAs was longer than distance from the incisors to the tip of the epiglottis, OPAs were partly withdrawn and repositioned the distal end of OPAs is placed just above the tip of epiglottis. Then, the length from the incisors to the flange of OPAs was measured. .

SUMMARY:
There are several studies that have measured various oropharyngeal airway space distances using radiological method. However, direct confirmation of optimal size of oropharyneal airways (OPAs) in individual using fiberoptic bronchoscope (FOB) is lacking as now. The purposes of this study were to directly determinate the proper size of OPA in individual by FOB via different sizes of OPA in adults under general anestheisia. Additionally, we examine the relationships among the size of OPA, straight length from the incisors to the tip of the epiglottis by laryngoscopy, patient height, and external facial measurements.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-II 2. 20-70 years adults

Exclusion Criteria:

* 1. an abnormal airway anatomy in preoperative radiologic study.
* 2. cervical spine pathology,
* 3. a history of difficult intubation,
* 4. neurologic disease or cardiovascular disease,
* 5. obesity (body mass index ≥ 30 kg m-1),
* 6. dental problem

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Optimal size of OPA | 1 min after each FOB measurement
  Primary Outcome - 기술(Description) The distance from the distal end of OPA to the tip of the epiglottis was calculated by the difference between measured distance from the incisors to the tip of the epiglottis via each OPA by FOB and typical distance from the flange to distal end of each OPA via inside tube of OPA. When the size of OPAs was longer than distance from the incisors to the tip of the epiglottis, OPAs were partly withdrawn and repositioned the distal end of OPAs is placed just above the tip of epiglottis. Then, the length from the incisors to the flange of OPAs was measured. The optimal size of OPAs in individuals was defined that the distal end of OPA is placed the tip of epiglottis as close as possible without impingement on the epiglottis when the flange of OPA contact with the four central incisors.

CONTACTS AND LOCATIONS:
Locations (1):
- Wyun Kon Park, Yonsei University College of Medicine, Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea